CLINICAL TRIAL: NCT01161173
Title: A Non-interventional Study to Follow and Evaluate Patients With Advanced NSCLC Who Are Treated in Second Line Setting With Tarceva (Erlotinib) in a "Real Life" Clinical Setting
Brief Title: An Observational Study of Tarceva (Erlotinib) in Routine Daily Clinical Practice as Second Line Treatment in Patients With Non-small Cell Lung Cancer
Acronym: TEAM
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21474
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Nonsquamous Nonsmall Cell Neoplasm of Lung
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Erlotinib: Participants received erlotinib (Tarceva) at a dose determined by the investigator, guided by the recommendation in the Summary of Product Characteristics. The recommended daily dose of erlotinib is 150 mg orally once daily.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib was provided in the retail versions of the product.
  Other Names: Tarceva

SUMMARY:
This observational study will evaluate the safety and efficacy of Tarceva (erlotinib) in routine clinical practice as second-line treatment in patients with recurrent or metastatic non-small dell lung cancer (NSCLC). Data will be collected from patients who have received 1 course of standard systemic chemotherapy, experienced disease progression, and who are receiveingTarceva in a second-line setting. Patients will also be followed through third-line treatment if there is disease progression on Tarceva therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Written informed consent.
* Recurrent or metastatic, Stage III or IV non-small cell lung cancer (NSCLC).
* Measurable disease (Response Evaluation Criteria In Solid Tumors).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Prior course of standard systemic chemotherapy.

Exclusion Criteria:

- Contra-indications to treatment with Tarceva.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients with progressive disease after first-line chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2008-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Belgium (30):
  - Aalst
  - Antwerp
  - Arlon
  - Bonheiden
  - Bouge
  - Boussu
  - Brussels
  - Charleroi
  - Chimay
  - Duffel
  - Edegem
  - Frameries
  - Genk
  - Gilly
  - Hasselt
  - Leuven
  - Liège
  - Marche-en-Famenne
  - Mons
  - Namur
  - Ostend
  - Ottignies
  - Roeselare
  - Seraing
  - Sint-Niklaas
  - Tournai
  - Turnhout
  - Verviers
  - Vilvoorde
  - Wilrijk
- Luxembourg (3):
  - Differdange
  - Esch-alzette
  - Luxembourg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 347
Completed | 0
Not Completed | 347
Not completed — Protocol Violation | 13
Not completed — Lost to Follow-up | 7
Not completed — Progressive Disease | 82
Not completed — Withdrawal of Consent | 5
Not completed — Unacceptable Toxicity | 21
Not completed — Death | 194
Not completed — End of Study | 2
Not completed — Reasons Not Specified | 23

BASELINE CHARACTERISTICS:
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol.
Groups:
- Cohort: Participants in the observational cohort received second-line therapy with Tarceva. At the time of discontinuation of Tarceva, a third-line chemotherapy or best supportive care were initiated as appropriate.
Arm/Group | Cohort
Number analyzed (Participants) | 334
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 239

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)
Description: The best overall response to treatment was determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. A CR was defined as the disappearance of all target lesions (TL) or the disappearance of all non-TLs. A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD. SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since treatment started for TLs and the persistence of 1 or more non-TL(s). PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs. For the best overall responses of CR and PR, a response was "confirmed" if a subsequent RECIST evaluation also showed a CR or PR.
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol. Only participants with an evaluable response were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 249
Percentage of participants
  Complete response | 0.8 [0.1 to 2.9]
  Partial response | 3.7 [1.7 to 6.9]
  Stable disease | 48.2 [41.7 to 54.6]
  Progressive disease | 47.3 [41.0 to 53.8]

2. Secondary Outcome: Time to Disease Progression
Description: The time to disease progression was defined as the time from Baseline until disease progression as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib
Number analyzed (Participants) | 334
Months | 3.6 [3.0 to 4.4]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from Baseline until disease progression or death from any cause. Progressive disease was determined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib
Number analyzed (Participants) | 334
Months | 2.7 [2.5 to 3.0]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from Baseline until or death from any cause
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib
Number analyzed (Participants) | 334
Months | 7.1 [5.1 to 9.5]

5. Secondary Outcome: Change From Baseline in the Lung Cancer Symptom Scale (LCSS) Scores
Description: Study participants and treating physicians completed the LCSS, a measure of Quality of Life (QoL), at Baseline and throughout the study. The patient LCSS measures 6 major symptoms, the Symptom Burden Index (SBI), associated with lung malignancies (3 thoracic [cough, dyspnea, haemoptysis] and 3 general symptoms [loss of appetite, fatigue, pain]) and 3 additional scores (overall symptomatic distress, interference with daily activities, global QoL), each on a 100 mm visual analogue scale (0=no impairment, 100=maximum impairment). The physician LCSS evaluates the 6 lung malignancy associated symptoms, the SBI, on an ordinal scale (100=none, 75=mild, 50=moderate, 25=marked, 0=severe). The average of the patient and physician SBI scores (6 symptoms) and the average of the patient total score (9 symptoms) ranged from 0 to 100, with a higher patient and a lower physician score indicating more impairment. A negative patient and a positive physician change score indicates improvement.
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol. Only participants with LCSS scores were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Erlotinib
Number analyzed (Participants) | 298
Units on a scale
  Patient SBI (n=283) | 0.15 [0.003 to 0.306]
  Patient total score (n=283) | 0.20 [0.020 to 0.370]
  Physician SBI (n=298) | -0.09 [-0.210 to -0.021]

6. Secondary Outcome: Percentage of Participants Who Developed Rash
Description: At each study visit, the presence of skin rash was graded using the Common Toxicity Criteria (CTC), with grade 0 = no rash, grade 1 = mild, grade 2 = moderate, grade 3 = severe, and grade 4 = life threatening or disabling rash. Reported is the percentage of participants who developed a grade ≥ 1 rash.
Time Frame: Baseline to the end of the study (up to 4 years, 4 months)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 334
Percentage of participants | 63.5 [58.0 to 69.0]

ADVERSE EVENTS:
Description: Safety analysis population: All participants who received at least 1 dose of erlotinib.
  The seriousness of adverse events was not captured in this observational study, therefore, all adverse events are reported as serious adverse events.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 210/347
Other Adverse Events (participants affected / at risk) | 0/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=347)
Death (General disorders) | 19 (19)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 16 (16)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Disease progression (General disorders) | 85 (85)
Fatigue (General disorders) | 4 (4)
General physical health deterioration (General disorders) | 19 (19)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Listeria sepsis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
General physical condition abnormal (Investigations) | 4 (4)
Liver function test abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Coma (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (3)
Loss of consciousness (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 18 (18)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights